CLINICAL TRIAL: NCT04662905
Title: A Prospective, Multicentre, Single-arm Feasibility Study Examining Novel Treatment Delivery of the Evoke Spinal Cord Stimulator (SCS) System to Treat Patients With Chronic Pain of the Trunk and/or Limbs
Brief Title: Novel Treatment Delivery of ECAP-controlled Closed-loop SCS for Chronic Pain
Acronym: Freshwater
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saluda Medical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-PCL-007873
Record Dates: First submitted 2020-11-30; First posted 2020-12-10 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Spinal Cord Stimulation; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ECAP-controlled, closed-loop SCS (Experimental): Spinal cord stimulation that measures and records evoked compound action potentials (ECAPs) and automatically adjusts the stimulation current to maintain a consistent ECAP amplitude
  Interventions: Device: Evoke Spinal Cord Stimulation (SCS) System

INTERVENTIONS:
Device: Evoke Spinal Cord Stimulation (SCS) System — ECAP-controlled, closed-loop SCS

SUMMARY:
The purpose of this study is to test and evaluate novel treatment delivery of ECAP-controlled closed loop SCS through the incorporation of new software and/or hardware features for patients with the Evoke System.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject has undergone trial implant or is planning to be implanted with the Evoke System within its approved indication.
* 2. Subject is willing and capable of giving informed consent and able to comply with study-related requirements.

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Evoke Compound Action Potentials (ECAPs) as measured by the Evoke SCS System | Through study completion, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Leitner, Study Director — Saluda Medical Pty Ltd
Locations (23):
- Australia (23):
  - ACT Pain Centre, Garran, Australian Capital Territory
  - Sydney Pain Specialists, Bella Vista, New South Wales
  - Genesis Research Services, Broadmeadow, New South Wales
  - Northern Integrated Pain Management, Charlestown, New South Wales
  - Australian Medical Research, Hurstville, New South Wales
  - Inner West Pain Centre, Newtown, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Northern Pain Centre, St Leonards, New South Wales
  - Women's Health & Research Institute of Australia, Sydney, New South Wales
  - Sydney Pain Research Centre Pty Ltd, Wahroonga, New South Wales
  - Interventus Pain Specialists, Auchenflower, Queensland
  - Axxon Pain Medicine, Brisbane, Queensland
  - Total Pain Clinic, Brisbane, Queensland
  - QPAIN, Fortitude Valley, Queensland
  - Sunshine Coast Clinical Research, Noosa, Queensland
  - Paul Frank Medical Services, Peregian Beach, Queensland
  - CerCare Pty Ltd, Wayville, South Australia
  - Monash Clinical Research, Clayton, Victoria
  - Frankston Pain Management, Frankston, Victoria
  - Pain Matrix, Geelong, Victoria
  - Melbourne Pain Specialists, Richmond, Victoria
  - Pain Specialists Australia, Richmond, Victoria
  - PainCare Perth, Cottesloe, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parker DJ, Antony AB, Smith GL, Goree JH, Russo MA, Petersen EA, Vu CM, Verrills P, Gilmore C, Kapural L, Nanavati D, Karantonis DM, Pope JE. Next-Generation SCS Programming Platform: Enhancing ECAP Fidelity and Objectivity to Improve Patient Experience. Pain Ther. 2026 Jan 8. doi: 10.1007/s40122-025-00808-5. Online ahead of print. PMID 41505067